CLINICAL TRIAL: NCT03796559
Title: A Prospective Open Label Study of the Use of Magseed® Markers and Sentimag® to Localize Axillary Lymph Nodes with Biopsy-proven Metastases in Breast Cancer Patients
Brief Title: Magseed Enabled Long-Term Localization of Axillary Lymph Nodes
Acronym: MAGELLAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endomagnetics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-003
Record Dates: First submitted 2018-11-08; First posted 2019-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Axillary Lymph Nodes
Keywords: Neo-adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Magseed marker (Experimental): Magseed marker deployed percutaneously, prior to patient undergoing neo-adjuvant chemotherapy (NAC), under ultrasound guidance to mark a lymph node intended for selective surgical removal post NAC.
  Interventions: Device: Magseed Marker

INTERVENTIONS:
Device: Magseed Marker — Implantable Magseed marker for marking lesions in soft tissue, detected using the Sentimag handheld probe.

SUMMARY:
The purpose of this study is to provide prospective evidence that the use of Magseed/Sentimag in marking axillary lymph nodes and guiding surgical localization in patients with breast cancer following neo-adjuvant chemotherapy (NAC) is effective.

DETAILED DESCRIPTION:
This is a post-market, prospective, open-label, single arm study of Magseed and Sentimag in patients with breast cancer with biopsy-proven axillary node metastases who had a clip placed to mark the metastatic node and are having that clipped node selectively removed at surgery following neo-adjuvant chemotherapy (NAC). Subjects will have the Magseed placed to mark axillary lymph nodes with biopsy-proven metastasis under ultrasound guidance before initiating NAC. After completion of NAC, the Magseed will be localized using the Sentimag system during surgery and removed with the targeted lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at time of consent
* Histologically confirmed cT0-4, N1 breast cancer
* Axillary lymph node metastasis with pathologic confirmation by needle biopsy
* Clip placed in the sampled axillary lymph node before initiation of chemotherapy
* Planned for neo-adjuvant chemotherapy prior to surgical resection
* Eligible for targeted axillary dissection (defined as selective localization and removal of the clipped node and SLND) at the completion of neo-adjuvant chemotherapy
* ECOG performance status 0-2

Exclusion Criteria:

* Distant metastases
* Inflammatory breast cancer
* Prior ipsilateral axillary surgical procedure including SLND or axillary node excision
* Prior history of breast cancer in the ipsilateral breast
* History of lymphoma
* Subject is pregnant
* Previous radiation to the breast or axilla
* Pacemaker or other implantable cardiac device in the ipsilateral chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Retrieval rate of clipped node and Magseed in the excised specimen | Time of surgery
  The retrieval rate of the clipped node and Magseed in the excised specimen. This is defined as the number of subjects in whom the clipped node and Magseed are retrieved in a single excised specimen divided by the total number of subjects.

SECONDARY OUTCOMES:
Rates of device and serious device-related events | Up to 42 days post-surgery
  Rates of device-related adverse events and serious device-related adverse events
Radiologic rated ease of Magseed placement | Time of Magseed marker placement
  5 point Likert scale, very easy = 5, very difficult = 1
Radiologic placement accuracy | Between completion of NAC time of surgery
  Success rate of seed placement (placement accuracy)
Radiologic seed position | After completion of NAC
  Success rate of maintained seed position at the completion of NAC
Surgical nodes localized | Time of surgery
  Number of nodes retrieved within the surgical specimen containing the Magseed
Ease of surgical localization | Time of surgery
  5 point Likert scalevery easy = 5, very difficult = 1

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Caudle, MD, MS, Principal Investigator — MD Anderson Cancer Center, Houston, TX
Locations (2):
- United States (2):
  - Baylor Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No